CLINICAL TRIAL: NCT00848146
Title: Natural Orifice Translumenal Endoscopic Surgery (NOTES)-Assisted Laparoscopic Cholecystectomy Surgery
Brief Title: NOTES-Assisted Laparoscopic Cholecystectomy Surgery
Acronym: TAS-NOTES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Principal Investigator, Eric Hungness, Assistant professor of surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23522; NU IRB# 1452-006
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Cholecystectomy, Laparoscopic; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NOTES-Assisted Lap Chole (Experimental): These patients will undergo an experimental surgical procedure that uses a combination of laparoscopic instruments (i.e., inserted through the skin into the abdominal cavity) and flexible endoscopic instruments (i.e., inserted through the mouth).
  Interventions: Procedure: Endoscopically assisted Laparoscopic Cholecystectomy Surgery

INTERVENTIONS:
Procedure: Endoscopically assisted Laparoscopic Cholecystectomy Surgery — Using endoscopic instruments a small incision will be made in the gastric wall and the endoscope will be advanced into the insufflated peritoneal cavity. At least one laparoscopic trocars will be placed through the abdominal wall for laparoscopic instrument insertion to manipulate and cut tissue. The flexible endoscope will provide visualization of the surgical field and flexible endoscopic instruments may be used to augment surgical manipulation with the laparoscopic instruments. The gallbladder will be removed through the stomach and out of the mouth. Endoscopic clips, sutures or tissue anchors (TAS)will be used to close the gastrotomy.
  Other Names: NOTES; Natural orifice translumenal endoscopic surgery; Transgastric Cholecystectomy

SUMMARY:
Refinements in laparoscopic surgery, coupled with advancements in therapeutic flexible endoscopy, have set the stage for surgery to move to even less invasive techniques to treat conditions in the GI tract and peritoneal cavity. Natural orifice translumenal endoscopic surgery (NOTES) offers a means of reducing and ultimately eliminating the need for abdominal incisions to gain access to the peritoneal cavity. In NOTES, a flexible endoscope and accessory instruments are inserted through a natural body orifice and passed through the wall of an organ to reach the abdominal cavity. By reducing or eliminating the need for abdominal incisions, NOTES may provide a least invasive surgical option that can reduce pain, recovery time, complications, and systemic inflammatory response when compared to a laparoscopic surgical approach. In this study, we propose to use the NOTES technique to eliminate the need for a 1.5-2.5 cm umbilical incision.

Hypothesis 1: We hypothesize that a combined endoscopic and laparoscopic approach will be able to eliminate a 1.5 to 2.5 cm infraumbilical incision when performing a laparoscopic cholecystectomy.

Hypothesis 2: Closure of the gastrotomy will be facilitated with the Ethicon TAS system.

DETAILED DESCRIPTION:
In this study, we propose to use a surgical technique that eliminates the need for a 1.5-2.5 cm umbilical incision. All patients will receive pre-operative antibiotics. A Veress needle will be used to create pneumoperitoneum with insufflation of carbon dioxide gas by a standard laparoscopic insufflator. A 5 mm laparoscopic port will be inserted through the abdominal wall in the right mid-abdomen and a 5 mm laparoscope inserted for viewing the abdominal cavity. A flexible endoscope, positioned within a multi-lumen 18 mm therapeutic access device, will be inserted through the mouth and into the stomach. Using commercially available endoscopes, endoscopic instruments and accessories, a small incision will be made in the gastric wall and the endoscope will be advanced into the insufflated peritoneal cavity. Additional laparoscopic trocars may be placed through the abdominal wall for laparoscopic instrument insertion to manipulate, retract and cut tissue. The flexible endoscope will provide visualization of the surgical field and flexible endoscopic instruments may be used to augment surgical manipulation with the laparoscopic instruments. Intraoperative cholangiogram or laparoscopic ultrasound will be performed at the discretion of the surgeon. Once dissected free, the gallbladder will be removed through the stomach and out of the mouth with the aid of an endoscopic retrieval bag. Commercially available endoscopic clips, or FDA approved tissue anchors will be used to close the gastrotomy. Additionally, the gastrotomy closure will be tested for leaks and laparoscopically oversewn with suture.

Operative and recovery room times as well as hospital length of stay will be collected. During the hospital stay, severity of pain, use of pain medications and complications will be recorded. Patients will be discharged per the standard of practice for a laparoscopic cholecystectomy. All study patients will receive a call from a surgery clinic nurse on post-op day 2 and 7. We will develop a check list that will contain the following (yes/no) elements to be used prior to discharge, on the post-op day 2 and 7 phone calls, and the 2 week post-op clinic visit: pain controlled with meds, nausea, emesis, fever, chills, redness of incisions, drainage from incisions, shortness of breath, chest pain, yellow eyes, dark urine, clay-colored stools. If there are any "yes" responses to this checklist prior to discharge, the patient will not be discharged from the hospital. If there are any "yes" responses to this checklist at the post-op day 2 or 7 phone call, the patient will be advised to immediately come to the GI surgery clinic or go to the nearest emergency room. If there are any "yes" responses to this checklist at the 2 week clinic visit, the patient will undergo the necessary standard of care medical evaluation (labs, tests, etc.) and may be admitted to the hospital. These checklists will be reviewed by one of the investigators, collected and stored in a locked file cabinet.

Patients will return and be evaluated by their surgeon two weeks following their procedure. At this visit, any post-operative complications will be noted in the patient's medical record. Additionally at this visit and at the preoperative visit, patients will complete a standardized Quality of Life (QOL) assessment (i.e., SF-36). Perceived pain levels and type and frequency of pain medications will be recorded in the patient's medical record.

The potential advantages to the patients entered into this study include those mentioned above regarding elimination of post-operative wound infection and hernia but also the lack of abdominal incisions greater than 5 mm in length may reduce pain and recovery time and likely have a cosmetic advantage as well. Potential risks of this study involve the risks of the standard laparoscopic procedure including bleeding, infection, injury to surrounding structures and port/trocar site pain. Potential risks associated with use of flexible endoscopic instruments include esophageal perforation, bleeding and sore throat. In addition, there is the possibility that there may be new, unanticipated complications from this modified surgical technique. Patient risks will be mitigated by having the procedure performed by a surgeon with expertise in both laparoscopic surgery and flexible endoscopy, as well as having involvement of a skilled interventional gastroenterologist if deemed necessary.

This feasibility study will initially evaluate the potential benefit, risks and impact on the patient's quality of life of this modified surgical technique in 10 patients. Once a standardized technique is established and risks are shown to be low, a prospective comparative evaluation is planned to compare this modified technique to the standard laparoscopic approach.

ELIGIBILITY:
Inclusion Criteria:

* Ability to undergo general anesthesia
* Age > 18 yrs. of age and < 85 yrs. of age
* Ability to give informed consent

Exclusion Criteria:

* Acute cholecystitis
* BMI > 40
* Contraindicated for esophagogastroduodenoscopy (EGD)
* Presence of common duct stones
* Presence of esophageal stricture
* Altered gastric anatomy
* Gallstone greater than 1.5cm diameter seen on pre-op ultrasound
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
post operative pain | two weeks

SECONDARY OUTCOMES:
quality of life | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Hungness, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States